CLINICAL TRIAL: NCT06740786
Title: Efficacy and Safety of Dapagliflozin in Preventing Atrial Fibrillation Recurrence After Catheter Ablation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Liu (Other)
Collaborators: Hefei Binhu Hospital (Other); The First People's Hospital of Hefei (Other); Second People's Hospital of Hefei City (Other); The Second People's Hospital of Anhui Province (Other)
Responsible Party: Sponsor-Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPAF
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): This group of patients will receive placebo treatment.
  Interventions: Drug: Dapagliflozin Treatment Group
- treatment group (Experimental): Dapagliflozin will be administered orally once daily at the recommended dose (e.g., 10 mg/day).
  Interventions: Drug: Dapagliflozin Treatment Group

INTERVENTIONS:
Drug: Dapagliflozin Treatment Group — This group of patients will receive dapagliflozin treatment after undergoing atrial fibrillation catheter ablation.
  Treatment regimen: Dapagliflozin will be administered orally once daily at the recommended dose (e.g., 10 mg/day).

SUMMARY:
Atrial fibrillation (AF) is a common arrhythmia, particularly prevalent in the elderly population. Catheter ablation is a common treatment for AF, but post-ablation recurrence of arrhythmias remains a significant clinical challenge. Dapagliflozin, an SGLT2 inhibitor primarily used for the treatment of type 2 diabetes, has shown potential in the field of cardiology, particularly for treating heart failure patients. Some studies suggest that dapagliflozin may reduce cardiac workload, improve heart function, and could even help in the management of atrial fibrillation. Therefore, this study aims to explore whether dapagliflozin can reduce the recurrence of arrhythmias following atrial fibrillation catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

- Age: Patients aged 18 years and older. Presence of type 2 diabetes or heart failure. Diagnosis of Atrial Fibrillation: Confirmed atrial fibrillation through ECG or Holter monitoring.

First-time Catheter Ablation: Patients undergoing their first atrial fibrillation catheter ablation.

Voluntary Participation: Patients willing to participate and sign informed consent.

Exclusion Criteria:

- Presence of urinary tract infection Pregnancy or Breastfeeding: Women who are pregnant, breastfeeding, or planning to become pregnant.

Allergy to Dapagliflozin or Similar Drugs: History of allergic reactions to dapagliflozin or other SGLT2 inhibitors.

Other Contraindications to Dapagliflozin: Any other contraindications for dapagliflozin use.

Kidney Function: eGFR < 45 ml/min/1.73m², with severe kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The recurrence of atrial arrhythmias | Within 12 months, beyond the 3-month blanking period.
  The recurrence of atrial arrhythmias within 12 months as assessed by ECG and holter, beyond the 3-month blanking period.

SECONDARY OUTCOMES:
The recurrence of atrial fibrillation | Within 12 months, beyond the 3-month blanking period.
  The recurrence of atrial fibrillation within 12 months as assessed by ECG and holter, beyond the 3-month blanking period.
changes in quality of life at 12 months as assessed by Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire | 12 months post-ablation.
  Quality of life was assessed using the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire, measuring changes from baseline to 12 months post-ablation.
Atrial Fibrillation Burden | after 1 year post-ablation
  Atrial fibrillation burden is defined as the percentage of time spent in atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) detected by a 7-day single-lead ECG patch monitoring after 1 year post-ablation.
Number of participants with adverse events | 12 months post-ablation.
  The safety of dapagliflozin assessed by researchers, including hypoglycemia, Urinary Tract Infections, dehydration and Hypotension,Acute Kidney Injury, diabetic ketoacidosi, cardiovascular events, severe allergic reactions, severe electrolyte Imbalance,etc.

IPD SHARING:
Plan to Share IPD: No